CLINICAL TRIAL: NCT03377582
Title: Virtual Reality Based-therapy Applied to Physical Therapy in Cardiology.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Ana Laura Ricci-Vitor, PhD, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCT400579/2017-0
Record Dates: First submitted 2017-11-06; First posted 2017-12-19 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Cardiac Disease; Risk Factor, Cardiovascular
Keywords: cardiovascular diseases; cardiac rehabilitation; sympathetic nervous system; heart rate; blood pressure; clinical trial; virtual reality exposure therapy; barriers to cardiac rehabilitation; motivation; adherence patient; engagement; perceived exertion; oxygen saturation
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Patient Compliance | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional therapy (Active Comparator): Exercise-based cardiac rehabilitation
  Interventions: Other: Exercise
- Virtual reality based therapy (Experimental): Exercise-based virtual reality
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Both interventions uses exercises

SUMMARY:
The aim of this study is to investigate engagement, motivation, and the barriers to adherence of virtual reality based therapy (VRBT) in patients with cardiac diseases and risk factors to the development of cardiac diseases. In addition, to investigate autonomic and hemodynamic responses of VRBT in comparison with conventional therapy (CT). To do this, patients with cardiac diseases or risk factors will be invited to perform CT or VRBT+CT. They will be submitted to an initial evaluation, and then will be random allocated to 12 weeks of intervention and to a final evaluation. The primary outcomes includes engagement, motivation, barriers and adherence in the 12 previous weeks using questionnaire, after 12 weeks of the intervention and after 12 weeks of the final intervention program. Hemodynamic and autonomic responses will be considered the secondary outcomes being evaluated before, during and after a session at the first, sixth and twelfth week.

DETAILED DESCRIPTION:
Introduction: cardiovascular rehabilitation programs (CR) can promote several benefits in patients with cardiac diseases. However, there are problems related to the patient adherence in CR. Some of these problems can be caused to factors like motivation. Alternative therapies can improve motivation and increase adherence to CR. In this context, virtual reality based therapy (VRBT), have shown benefits in cardiac patients to pain relief, functional capacity and increasing physical activity levels, but there is no answer whether it can increase engagement and adherence to CR. In addition, it is important to investigate hemodynamic responses of VRBT. Objective: investigate engagement, motivation, and the barriers to adherence of VRBT in patients with cardiac diseases and risk factors to the development of cardiac diseases. In addition, to investigate autonomic and hemodynamic responses of VRBT in comparison with conventional therapy (CT). Methods: patients with cardiac diseases or risk factors will be invited to perform CT or VRBT+CT. They will be submitted to an initial evaluation, the intervention and to a final evaluation. The initial evaluation include eligibility investigation, and after they will be random allocated to the interventions. The interventions will be performed with a frequency of three times a week, for 12 weeks, and the intensity will be prescribed individually. The primary outcomes includes engagement, motivation, barriers and adherence in the 12 previous weeks according to a recall questionnaire, after 12 weeks of the intervention and after 12 weeks of the final intervention program. The engagement will be evaluated using the User Engagement Scale (modified). Motivation will be evaluated using the intrinsic motivation questionnaire. The barriers will be evaluated using the Barriers Scale of Cardiac Rehabilitation. Adherence will be evaluated using the presence in the patient's records. Hemodynamic responses will be evaluated before, during and after a session at the first, sixth and twelfth week using blood pressure, heart rate, respiratory rate, oxygen saturation and rating of perceived exertion. Autonomic responses will be evaluated using heart rate variability. Statistical analysis: the data analysis will be evaluated using the two way ANOVA with Bonferroni posttest with significance to p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cardiovascular diseases
* Patients with risk factors to develop cardiovascular diseases

Exclusion Criteria:

- Patients who disagree to participate of any protocol interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Engagement | Change from baseline at 12 weeks
  Measured using the Utrecht engagement scale modified There is 17 items scored from 1 to 7, according to the Likert Scale. Then, each item is summed and divided for the number of items. Higher values represent a better engagement.
Motivation | Change from baseline at 12 weeks
  Measured using the Intrinsic motivation inventory There is 18 items scored from 1 to 5, according to the Likert Scale. Then, each item is summed and divided for the number of items. Higher values represent a better motivation.
Barriers to Cardiac Rehabilitation | Change from baseline at 12 weeks
  Measured using Cardiac Rehabilitation Barriers Scale There is 21 items score from 1 to 5, according to the Likert Scale. Then, each item is summed and divided for the number of items. Higher values represent a worse outcome. In addition, there is four subscales: 1) Perceived need/health care factors, 2) Logistical factors, 3) Work/time conflicts, and 4) Comorbidities/functional status. The subscales are scored in the same way of the total, it means, from 1 to 5 and them dividing from the total number of the items included in the subscale.
Adherence to Cardiac Rehabilitation | Change from baseline at 12 weeks
  Measured using the number of cardiac rehabilitation sessions attended

SECONDARY OUTCOMES:
Autonomic responses | Up to 12 weeks
  Measured using heart rate variability The heart rate variability will be measured through the following linear indices (SDNN: the standard deviation of normal-to-normal intervals, ms; rMSSD: the root mean square of successive difference between normal intervals,ms; RRtri: triangular index, based on RR intervals,ms; TINN: triangular interpolation of the normal to normal interval between consecutive heart beats, ms; LF: low frequency, nu; HF: high frequency and nonlinear indices,nu.). In addition the nonlinear indices will be measured (SD1: standard deviation of instant variability beat to beat; SD2: standard deviation of long-term interval between consecutive heart beats). In general higher values represent a better autonomic response.
Blood pressure | Up to 12 weeks
  Measured using both systolic blood pressure and diastolic blood pressure
Heart rate | Up to 12 weeks
  Measured using an equipment validated for recording heart rate beat to beat
Respiratory rate | Up to 12 weeks
  Measured using the number of respiratory incursions in one minute
Oxygen Saturation | Up to 12 weeks
  Measured using an oximeter
Perceived exertion | Up to 12 weeks
  Measured using Borg Scale. This scale varies from 6 to 20.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Laura Ricci-Vitor, PhD, Principal Investigator — Universidade Estadual Paulista Júlio de Mesquita Filho
Locations (1):
- Laboratório de Fisiologia do Estresse, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
After published results,

REFERENCES:
- [Derived] da Cruz MMA, Ricci-Vitor AL, Borges GLB, da Silva PF, Turri-Silva N, Takahashi C, Grace SL, Vanderlei LCM. A Randomized, Controlled, Crossover Trial of Virtual Reality in Maintenance Cardiovascular Rehabilitation in a Low-Resource Setting: Impact on Adherence, Motivation, and Engagement. Phys Ther. 2021 May 4;101(5):pzab071. doi: 10.1093/ptj/pzab071. PMID 33625515
- [Derived] Alves da Cruz MM, Ricci-Vitor AL, Bonini Borges GL, Fernanda da Silva P, Ribeiro F, Marques Vanderlei LC. Acute Hemodynamic Effects of Virtual Reality-Based Therapy in Patients of Cardiovascular Rehabilitation: A Cluster Randomized Crossover Trial. Arch Phys Med Rehabil. 2020 Apr;101(4):642-649. doi: 10.1016/j.apmr.2019.12.006. Epub 2020 Jan 8. PMID 31926142